CLINICAL TRIAL: NCT00426036
Title: An Open-Label Study in Healthy Subjects and in Patients With Stable Impaired Renal Function to Assess the Effect of Severe Renal Impairment on Licarbazepine Pharmacokinetics and Metabolism After the Single Administration of a 500 mg Licarbazepine Immediate Release (IR) Tablet
Brief Title: Effect of Severe Renal Impairment on Pharmacokinetics and Metabolism of a Single Administration of Licarbazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIC477D2311
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Open-label study, healthy subjects, stable impaired renal function, licarbazepine, pharmacokinetics, metabolism, safety.
MeSH Terms: interventions — 10,11-dihydro-10-hydroxy-5H-dibenz(b,f)azepine-5-carboxamide

INTERVENTIONS:
Drug: Licarbazepine

SUMMARY:
This study will assess the influence of severe renal impairment on the pharmacokinetics of licarbazepine and its glucuronide conjugate after single oral administration in healthy subjects and in subjects with stable impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects/patients from 18-60 years of age
* Body mass index (BMI) must be within the range of 18 and 30 kg/m². Subjects/patients must weigh a minimum of 50 kg.
* Female subjects/patients must either have been surgically sterilized or hysterectomized at least 6 months prior to screening.
* Subject/patient must be able to provide written informed consent prior to study participation.

Exclusion Criteria:

* Clinically significant abnormal laboratory values at the screening evaluation or at the baseline re-evaluation, for patients excluding those normally associated with severe degree of renal impairment or the primary cause of renal insufficiency.
* Use of any over-the-counter medications or herbal / natural supplements during 2 weeks prior to dosing. (acetaminophen is acceptable, but must be documented in the Concomitant Medications / Non-Drug Therapies page of the CRF).
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing or other amount considered to compromise the health of the subject/patient if previous history of anemia exists.
* Significant acute illness within the two weeks prior to dosing.
* History of any significant cardiovascular events (M.I., angioplasty, angina) within 6 months of study start.
* A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
* History of hyponatremia.
* History of seizures.
* Any surgical or medical condition which might significantly alter the absorption,distribution, metabolism or excretion of drugs other than renal impairment or which may jeopardize the subject/patient in case of participation in the study. The investigator should be guided by history of any of the following: inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding gastropathy (gastroparesis) or enteropathy major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection clinical evidence of pancreatic injury or pancreatitis
* History of immunocompromise, including a positive HIV (ELISA and Western blot) test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result .
* History of drug or alcohol abuse within the 6 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-06

PRIMARY OUTCOMES:
Influence of severe renal impairment on pharmacokinetics of
licarbazepine and its glucuronide conjugate after single oral dose of 500 mg licarbazepine IR in healthy subjects and in severe renal impaired patients.

SECONDARY OUTCOMES:
Influence of severe renal impairment on pharmacokinetics of two enantiomers of licarbazepine, the glucuronide conjugates of licarbazepine and its two enantiomers after single oral dose of 500 mg licarbazepine IR in healthy subjects and i
Safety and tolerability of single oral doses of 500 mg given as one 500 mg IR tablet in healthy subjects and in severe renal impaired patients.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis Investigative site, Prague, Czechia